CLINICAL TRIAL: NCT06207721
Title: Physical Therapy for Functional Constipation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Associated professor at faculty of physical therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: constipation in children
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Physical Therapy in Pediatric Functional Constipation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (A) (Experimental): conventional treatment by diet regimen and laxatives
  Interventions: Drug: Polyethylene Glycols
- study Group (B) (Experimental): physical therapy program in addition to conventional treatment by diet regimen and laxatives
  Interventions: Drug: Polyethylene Glycols; Other: Physical therapy program

INTERVENTIONS:
Drug: Polyethylene Glycols — Polyethylene Glycols syrup (0.7 g/kg daily)
Other: Physical therapy program — The physical therapy program includes exercises and massage
  Arms: study Group (B)

SUMMARY:
Children diagnosed with functional constipation are subjected to physical therapy combined with conventional treatment

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed as functional constipation.
* aged from 4 to 18 years old
* from both sex

Exclusion Criteria:

* children diagnosed as constipation caused by medicine Bowel surgery, Endocrine and metabolic disorders , Neurological and psychiatric disorders.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Rome-III criteria | after 6 months of interventions
  assessment for functional constipation symptoms

SECONDARY OUTCOMES:
short form 36 questionnaire | after 6 months of interventions
  assessment for quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

REFERENCES:
- [Derived] Soliman A, AboAli SEM, Abdel Karim AE, Elsamahy SA, Hasan J, Hassan BA, Mohammed AH. Effect of adding telerehabilitation home program to pharmaceutical treatment on the symptoms and the quality of life in children with functional constipation: a randomized controlled trial. Eur J Pediatr. 2024 Sep;183(9):3943-3958. doi: 10.1007/s00431-024-05639-8. Epub 2024 Jun 26. PMID 38922435